CLINICAL TRIAL: NCT01809223
Title: The Safety and Efficacy of Conbercept in the Treatment of Choroidal Neovascularization (CNV) Secondary to High Myopia
Brief Title: A Randomized, Double-blind, Multicenter, Sham-controlled, Safety and Efficacy Study of Conbercept in Patients With mCNV
Acronym: SHINY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHSWKH902007
Record Dates: First submitted 2013-03-11; First posted 2013-03-12 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-03

CONDITIONS: Choroid Neovascularization Secondary to Degenerative Myopia
MeSH Terms: interventions — KH902 fusion protein; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- conbercept treatment group (Experimental): Subjects will receive conbercept injections at a dose of 0.5 mg/eye, once a month for first 3 months. In the next 6 months, the investigator will decide whether repeat injections are needed base on the monthly assessment results.
  Interventions: Drug: conbercept, Fixed; Drug: conbercept, PRN
- sham injection group (Sham Comparator): Subjects will receive sham injections monthly for 3 months and will receive 0.5 mg/eye conbercept at month 4. The investigator will decide whether repeat injections are needed base on the monthly assessment results from month 5 to month 9.
  Interventions: Drug: conbercept, Fixed; Drug: conbercept, PRN; Other: sham injection

INTERVENTIONS:
Drug: conbercept, Fixed — intravitreal injection of 0.5 mg conbercept per month, fixed injection
Drug: conbercept, PRN — intravitreal injection of 0.5 mg conbercept as need, PRN
Other: sham injection — sham intravitreal injection per month, fixed injection
  Arms: sham injection group

SUMMARY:
This study is design to evaluate the effect of conbercept therapy on visual acuity and anatomic outcomes compared to sham injection and durability of response observed in subjects with choroid neovascularization secondary to pathological myopia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients give fully informed consent and are willing and able to comply with all study procedures.
2. In the study eye:

   * Myopia of equal to or greater than -6.00D,and axial length ≥26.5mm.
   * Diagnosis of active subfoveal, juxafoveal, or extrafoveal CNV secondary to high myopia.
   * Visual impairment due to CNV secondary to high myopia.
   * BCVA score ≥24 and ≤73 ETDRS letters (approximately 20/40~ 20/320 Snellen equivalent).
   * Ocular media of sufficient quality to obtain fundus and OCT images.
3. The BCVA score of fellow eyes ≥ 19 ETDRS letters (approximately 20/400 Snellen equivalent)

Exclusion Criteria:

1. Current vitreous hemorrhage in either eye.
2. Intraocular treatment with corticosteroids within last 3 months or periocular treatment with corticosteroids within last month in the study eye.
3. Active infectious ocular inflammation in either eye.
4. Fibrosis or atrophy involving the center of foveal in the study eye.
5. Any concurrent intraocular condition in the study eye that, in the opinion of investigator, could either require medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition.
6. The lesion size ≥30 mm2 in the study eye.
7. Any ocular disorder in the study eye that, in the opinion of the investigator, may confound interpretation of the study results.
8. Uncontrolled glaucoma or cup/disk ratio > 0.8 in the study eye.
9. Aphakia (excluding artificial lens) in the study eye.
10. Serious amblyopia and amaurosis in the fellow eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
mean change from baseline of visual acuity | 3-month
  to compare the mean change from baseline of best-corrected visual acuity (BCVA) between conbercept treatment group and sham injection group at month 3

SECONDARY OUTCOMES:
mean change from baseline of anatomical features | 3-month
  to compare the difference of mean change from baseline of CRT, CNV size and lesion size between conbercept treatment group and sham injection group at month 3
mean change from baseline of visual acuity | 9 months
  to evaluate the mean change from baseline of BCVA of two groups from month 1 to month 9
safety and tolerability of conbercept | 3-month and 9-month
  to evaluate the incidence of AEs (ocular or non-ocular) of two groups at month 3 and 9

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tongren hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Daping Hospital, Research Institute of Surgery Third Military Medical University, Chongqing, Chongqing Municipality
  - Zhongshan Ophthalmic Center, Guangzhou, Guangdong
  - Wuhan General Hospital of Guangzhou Military, Wuhan, Hubei
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Ophthalmologic Hospital of Qingdao, Qingdao, Shandong
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xian, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Affiliated Eye Hospital of WMC, Wenzhou, Zhejiang